CLINICAL TRIAL: NCT04554758
Title: Korean OBEsity Surgical Treatment Study(KOBESS-II) : Protocol of a Prospective Multicenter Cohort Study on Morbid Obesity Patients Undergoing Sleeve Gastrectomy Versus Roux-en Y Gastric Bypass
Brief Title: Comparative Analysis Between Sleeve Gastrectomy and Roux-en Y Gastric Bypass in Bariatric Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Yoonseok Heo, Professor, Inha University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOBESS-II trial
Record Dates: First submitted 2020-09-09; First posted 2020-09-18 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Obesity, Morbid; Overnutrition; Nutrition Disorders; Overweight and Obesity; Body Weight Changes
Keywords: primary bariatric surgery; morbid obesity; sleeve gastrectomy; Roux-en Y gastric bypass; South Korea
MeSH Terms: conditions — Obesity, Morbid; Overnutrition; Nutrition Disorders; Overweight; Obesity; Body Weight Changes | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Comparative double arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve gastrectomy (Experimental): 200 obesity patients who undergo laparoscopic sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy
- Roux-en-Y gastric bypass (Experimental): 200 obesity patients who undergo laparoscopic Roux-en-Y gastric bypass
  Interventions: Procedure: Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Bariatric operation will be done by laparoscopic sleeve gastrectomy procedure.
  Arms: Sleeve gastrectomy
Procedure: Roux-en-Y gastric bypass — Bariatric operation will be done by laparoscopic Roux-en-Y gastric bypass procedure.
  Arms: Roux-en-Y gastric bypass

SUMMARY:
Prospective, double-arm, multi-center cohort study on obese patients, for laparoscopic sleeve gastrectomy versus Roux-en Y gastric bypass

DETAILED DESCRIPTION:
This is prospective cohort study. Total 400 obese patients will be enrolled(Sleeve gastrectomy 200 patients, Roux-en-Y gastric bypass 200)

The principal investigator or another clinical investigator in charge will individually inform the patients about the study, before operation at out patient clinic. At that time patient is selected to either sleeve gastrectomy group or Roux-en-Y gastric bypass group. All investigator report to clinical research center about patients BMI and operation method.

About 30-35 obesity patients will be enrolled according to their BMI status. Patients' BMI status is classified into several parts by 2.5 gap started from 27.5.

All patients will undergo periodically anthropometry, laboratory tests, bioelectrical impedance analysis, gastrofiberscopy, polysomnography and abdomen CT before and after surgery.

Patients with hypertension will undergo echocardiography. Patients with polycystic ovary syndrome will be checked hormonal study. Patients with type 2 diabetes mellitus will be performed 75g oral glucose tolerance test test.

Surgical complication include wound morbidities, gastrointestinal leakage or fistula, postoperative bleeding, intra-abdominal abscess, stricture , adhesive ileus, reflux esophagitis, marginal ulceration, dumping syndrome and internal hernia.

Systemic complication which is not associated with the operation field include ling morbidities, heart morbidities, urinary morbidities and others.

Hospital mortality is defined as postoperative death form any cause within 30 days after operation.

All patients will be followed up post operative 1 month, 3 month, 6 month, 12 month, 18 month, 24 month.

All patients' liver tissue, visceral fat and subcutaneous fat will be harvested during operation.

All patients' blood sample will be collected at out patient clinic visit. All patients' urine and face will be collected at out patient clinic visit and will be analyzed to evaluate microbial change throughout pre and post operation period.

ELIGIBILITY:
Inclusion Criteria:

* obesity patients(BMI over 35)
* morbid obesity patients(BMI over 30) with cardiovascular disease, hypertension, hyperlipidemia, type 2 diabetes mellitus, obstructive sleep apnea
* type 2 diabetes mellitus obesity patients(BMI over 27.5) who were treated medical therapy or HbA1C level over 7%

Exclusion Criteria:

* Patients who underwent previously bariatric operation
* Patients who were diagnosed malignant disease patients within 5 years
* Patients who were involved with other clinical trial within 3 months
* Patients who are risky to conduct general anesthesia for operation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Obesity Cure Success Rate | Postoperative 1 year
  Proportion of patients who reach BMI bellow 25
Body weight change rate | Postoperative 1 year
  Decreased body weight proportion compare to preoperative body weight
Waist circumference change rate | Postoperative 1 year
  Decreased waist circumference change proportion compare to preoperative waist circumference

SECONDARY OUTCOMES:
Rate of morbid disease remission or partial remission | Postoperative 1 year, 2 year
  Remission rate or partial remission rate of morbid disease related to obesity such as hypertension, type 2 diabetes mellitus, hyperlipidemia after surgery
Postoperative complication rate and mortality rate | Within postoperative 30 days
  Number of participants surgical complications associate with the surgical technique or the operation field Number of participants mortality after operation associated with surgical complication or underlying disease
Micronutrient deficiency | Postoperative 1 year, 2 year
  Incidence of micronutrient deficiency rate such as vitamine, calcium, iron
Quality of life improvement rate and degree-1 | Postoperative 1 year, 2 year
  Patients rate and quantitative analysis of the improved life quality using several survey EQ-5D-3L(EuroQol-5D) consists of 5 dimensions(mobility, self-care, usual activities, pain/discomfort and anxiety/depression).
  Each of which is scored as no/some/extreme problems. The dimension scores are converted into health utility scores ranging form 0(death) to 1(perfect health)
Quality of life improvement rate and degree-2 | Postoperative 1 year, 2 year
  EQ-VAS(EuroQol-Visual Analogue scale) is a question scale ranging form 0 to 100.
  0 indicated the worst and 100 indicated the best condition. EQ-VAS provides important, complementary information on patient's view about their own health.
Quality of life improvement rate and degree-3 | Postoperative 1 year, 2 year
  Impact of Weight on QoL(IWQoL) has 5 dimensions and each dimension has several items.
  * physical function : 11 items
  * self-esteem : 7 items
  * sexual life : 4 items
  * public distress : 5 items
  * work : 4 items
  Score range from 0 to 100 and 100 represents the best quality of life.
Quality of life improvement rate and degree-4 | Postoperative 1 year, 2 year
  Moore-head-Ardelt QoL questionnaire II(MA-II) has 6 items(general self-esteem, physical activity, social contacts, satisfaction concerning work, pleasure related to sexuality and focus on eating behavior).
  All items are scored according to 10-level Likert scale(-0.5 to 0.5) and all have the same weight.
Quality of life improvement rate and degree-5 | Postoperative 1 year, 2 year
  Obesity-related Psychosocial Problem scale(OP scale) consists of 8 items that measure the bothersome impact of body weight on given situations.
  (private gatherings in their own home, private gatherings at their friend or relative's home and going to restaurant)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Seok Heo, Professor, Principal Investigator — Inha University Hospital; Do Joong Park, Professor, Study Director — Seoul National University Hospital; Yong Suk Park, Professor, Study Director — Seoul National University Bundang Hospital; Seung Wan Ryu, Professor, Study Director — Keimyung University Hospital; Moon Won Yoo, Professor, Study Director — Ulsan univertisy Seoul Asan Medical Center; Han Hong Lee, Professor, Study Director — The Catholic University of Korea; Ji Yeon Park, Professor, Study Director — Kyungpook National University Hospital; Sang Hyun Kim, Professor, Study Director — Soonchunhyang University Hospital; Jong Won Kim, Professor, Study Director — Chung-Ang University Hopspital; Jong Han Kim, Professor, Study Director — Korea University Medical Center(Guro Hospital); In Seob Lee, Professor, Study Director — Ulsan univertisy Seoul Asan Medical Center; In Gyu Kwon, Professor, Study Director — Yonsei University Medical Center(Gangnam Hospital); Tae Kyung Ha, Professor, Study Director — Hanyang University; Sung Il Choi, Professor, Study Director — Kyung Hee University Hospital at Gangdong; Kyung Won Seo, Professor, Study Director — Kosin University Gospel Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea